CLINICAL TRIAL: NCT04803045
Title: The Impact of a Brief Intervention on Retention Rates With Patients Who Did Not Return to Care After an Initial Physician Visit
Brief Title: Does a Brief Intervention Decrease Patient Drop Out Rates?
Status: Completed | Type: Observational
Sponsor: Boston IVF (Other)
Responsible Party: Sponsor
Other Study IDs: DomarRTC
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Infertility
Keywords: Infertility; IVF; Patient retention
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Follow Up Email: Patients received a follow up email 3 months after an initial consult with a physician but did not return to care.
  Interventions: Other: Follow up email
- No follow up: Patients who did not receive any follow up after their initial consult, following clinic standard of care.

INTERVENTIONS:
Other: Follow up email — Patients received an email 3 months after an initial consult asking why they had not returned to care. Patients were provided with 4 options and a space to write in comments. The email asked if the patient had any questions and offered support.
  Groups: Follow Up Email

SUMMARY:
The goal of this study is to determine a) if a follow-up email to selected patients who had an initial consult with an infertility specialist, but did not return for a second visit, would change return to care behavior and b) why patients had not returned.

DETAILED DESCRIPTION:
From July 2017 to March 2018 all patients who had attended an initial visit with an infertility specialist at the clinic, but had not returned for at least three months were selected to receive a follow up email. Those selected for an email excluded patients who the Investigator's knew had achieved a pregnancy, already had a plan for treatment, had visited for an egg freeze and all LGTBQ patients. The email asked if the patient had any questions about that visit, offered support to the patient and included contact information for the patient liaison sending the email. The email also asked each participant to indicate why they had not returned and were provided 4 options and an opportunity to write in a response. From April 2018 to December 2018 no emails were sent to patients. No other change of patient contact practice was initiated during the trial period. This study will observe routine to care behavior of these patients after 11 months post initial consult date.

ELIGIBILITY:
Inclusion Criteria:

* Female patients attending an initial consult with a physician at Boston IVF and were recommended to continue care with the clinic

Exclusion Criteria:

* Patients who the Investigators knew had achieved a pregnancy
* Patients who already had a plan for treatment in place after their initial consult
* Patients who had visited for an egg freeze
* LGTBQ patients

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Female patients attending an initial consult at Boston IVF between set dates.
Sampling Method: Non-Probability Sample
Enrollment: 647 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Return to care behavior | 11 months after initial consult
  The study will track if the patient return to care rate

CONTACTS AND LOCATIONS:
Overall Officials: Alice Domar, PhD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No